CLINICAL TRIAL: NCT05172544
Title: A Double Blind, Randomized, Placebo-Controlled, Phase 1 Dose Escalation Trial to Evaluate the Safety and Immunogenicity of an Inactivated Yellow Fever Virus Vaccine, HydroVax-002 YFV, in Healthy Adults
Brief Title: Trial of an Inactivated Yellow Fever Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Najit Technologies, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20-001; 4U44AI145791-02 (NIH)
Record Dates: First submitted 2021-12-07; First posted 2021-12-29 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Yellow Fever
Keywords: HydroVax; Yellow Fever virus; dose-ranging; double blind; Placebo-Controlled; Vaccine
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose Sentinel (Experimental): 3 subjects will receive 1 mcg intramuscularly (IM) of HydroVax-002 YFV and 1 subject will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-002 YFV; Other: Placebo
- Low Dose Expanded (Experimental): 7 subjects will receive 1 mcg intramuscularly (IM) of HydroVax-002 YFV and 2 subject will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-002 YFV; Other: Placebo
- High Dose Sentinel (Experimental): 3 subjects will receive 5 mcg intramuscularly (IM) of HydroVax-002 YFV and 1 subject will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-002 YFV; Other: Placebo
- High Dose Expanded (Experimental): 7 subjects will receive 5 mcg intramuscularly (IM) of HydroVax-002 YFV and 1 subject will receive placebo IM on Days 1 and 29.
  Interventions: Biological: HydroVax-002 YFV; Other: Placebo

INTERVENTIONS:
Biological: HydroVax-002 YFV — Inactivated YFV vaccine
Other: Placebo — NaCl 0.9%, Normal Saline

SUMMARY:
This trial will be a randomized, placebo controlled, double-blind (within dosing group), dose escalation Phase 1 trial, evaluating dosages of 1 mcg and 5 mcg of HydroVax-002 YFV vaccine given intramuscularly on Day 1 and Day 29 in up to 25 healthy adults healthy adults ≥ 18 and < 50 years of age. The primary objective is to assess the safety, reactogenicity, and tolerability of the HydroVax-002 YFV vaccine administered intramuscularly in a two-dose series on Days 1 and 29 at a dose of 1 mcg or a dose of 5 mcg.

DETAILED DESCRIPTION:
This trial will be a randomized, placebo controlled, double-blind (within dosing group), dose escalation Phase 1 trial evaluating dosages of 1 mcg and 5 mcg of HydroVax-002 YFV vaccine given intramuscularly on Day 1 (the day of first vaccination is defined as Day 1) and Day 29 in healthy adults ≥ 18 and < 50 years of age. The study will consist of two dosing groups of HydroVax-002 YFV vaccine to be enrolled sequentially. Each dose group will consist of 10 individuals who receive HydroVax-002 YFV, as well as 5 total subjects who receive placebo. Each dose-group will include a sentinel subgroup consisting of 3 vaccine and 1 placebo recipient. In each of the two (1 mcg and 5 mcg) dose phases, enrollment is halted after the dose 1 vaccination of the sentinel subgroup. Following assessment of safety and reactogenicity data of Group 1 by the Safety Monitoring Committee (SMC), the vaccine dose will be increased to 5 mcg for Group 2.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Must agree to the collection of venous blood per protocol.
4. Are males or non-pregnant females, ≥18 and <50 years of age, inclusive at time of enrollment.
5. Are in good health*. *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, emergency room or urgent care for condition, or invasive medical procedure and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose or in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening or treatment of continued symptoms of medical diagnosis or condition. Note: Low dose topical, corticosteroids as outlined in the Subject Exclusion Criteria (see below) as well as herbals, vitamins and supplements are permitted.
6. Oral temperature is less than 100.0°F.
7. Pulse is 47 to 100 beats per minute, inclusive.
8. Systolic blood pressure is 85 to 140 mmHg, inclusive.
9. Diastolic blood pressure is 55 to 90 mmHg, inclusive.
10. Screening laboratories (WBC, Hgb, PLTs, Sodium, Potassium, Bicarbonate, Calcium, Cr, non-fasting glucose, ALT, AST, TBIL and urine protein and glucose) are within acceptable parameters*. *Hematology, blood chemistry and liver enzymes must be Grade 1 or less at screening; urine glucose and protein negative at screening for subjects to qualify for randomization and vaccination.
11. Negative test for HIV, hepatitis B virus (HBV), and hepatitis C virus (HCV) at screening blood draw.
12. Women of childbearing potential* must use an acceptable contraception method† from at least 30 days before the first study vaccination until 30 days after the second study vaccination. *Not sterilized via, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal. †Includes non-male sexual relationships, full abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more and shown to be azoospermic prior to the subject receiving the study vaccination, effective intrauterine devices, NuvaRing®, tubal ligation, and licensed hormonal methods such as implants, injectables or oral contraceptives (i.e. "the pill").
13. Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.
14. Sexually active males must agree to use a medically acceptable form of contraception* in order to be in this study and must agree to continue such use until day 30 after the last vaccination. *Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicide. Contraceptive measures such as Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.

Exclusion Criteria:

1. Have an acute illness* or acute febrile illness (oral temperature ≥ 38C [100.4F]), as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination. *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation*. *Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Known allergy to components of the study product*. *Including the following: aluminum hydroxide, sorbitol, potassium chloride, sodium chloride and polysorbate80 (Tween80)
7. Unstable seizure disorder (defined as requiring medication for seizure control or with seizure activity within the past 3 years).
8. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
9. Have any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere* with subject compliance or safety evaluations. *As determined by the site PI or appropriate sub-investigator.
10. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
11. Have a history of asthma, other than mild, well-controlled asthma*. *Cold or exercise induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Participants should be excluded if they require daily bronchodilator use, or have had an asthma exacerbation requiring oral/parenteral steroid use or have used theophylline or inhaled corticosteroids in the past year.
12. Have a history of diabetes mellitus.
13. Have taken oral or parenteral (including intra-articular) or chronic topical corticosteroids of any dose within 30 days prior to study vaccination*. *Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis may be enrolled the day after their therapy is completed.
14. Have taken high-dose inhaled corticosteroids* within 30 days prior to study vaccination. *High-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE.
15. Received or plan to receive a licensed, live vaccine within 30 days before or after each study vaccination.
16. Received or plan to receive a licensed, inactivated vaccine or allergy desensitization shot within 14 days before or after each study vaccination.
17. Received an experimental agent* within 30 days prior to the study vaccination or expect to receive another experimental agent† during the trial-reporting period‡. *Including vaccine, drug, biologic, device, blood product, or medication. †Other than from participation in this trial. ‡Approximately 7 months after the first study vaccination.
18. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the trial-reporting period†. *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication. †Approximately 7 months after the first study vaccination.
19. Female subjects who are breastfeeding or plan to breastfeed from the time of the first study vaccination through 30 days after the last study vaccination.
20. Receipt of blood products or immunoglobulin within six months prior to enrollment.
21. Donation of a unit of blood within 60 days prior to enrollment or intends to donate blood during the study period.
22. Body mass index (BMI) ≥ 35.
23. History of a visit to South America, sub-Saharan Africa or Southeast Asia lasting one month or more.
24. Planned travel to areas known to be endemic with Yellow Fever virus during the study period.
25. History of military service.
26. History of vaccination against dengue, yellow fever, tick-borne encephalitis, or Japanese encephalitis.
27. History of vaccination with other flavivirus candidate vaccines.
28. Attended primary (grade) school in Austria, Germany, Japan, South Korea, India, Thailand, Nepal, Vietnam, or Taiwan (locations where the tick-borne encephalitis vaccine is given).
29. History of yellow fever.
30. Plan to have a major change in exercise routine or perform strenuous exercise from 72 hours before any dose of study vaccine/placebo and for 72 hours before any safety laboratories*. *Safety laboratories are obtained on Days 4 and 15 following each dose of study product.
31. Contraindication to intramuscular vaccination of either upper arm (for example, due to lymphadenectomy or obscuring tattoos).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W Woods, MD, MPH, Principal Investigator — Duke Health; Emmanuel B Walter, MD, MPH, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose: 1 mcg intramuscularly (IM) of HydroVax-002 YFV on Days 1 and 29.
- High Dose: 5 mcg intramuscularly (IM) of HydroVax-002 YFV on Days 1 and 29.
- Placebo: Placebo intramuscularly (IM) on Days 1 and 29.
Period: Overall Study
Arm/Group | Low Dose | High Dose | Placebo
Started | 10 | 10 | 6 (Prior to receiving the first vaccination, one placebo subject was discontinued from the study by physician decision and was replaced.)
Completed | 9 (One subject voluntarily withdrew from the study prior to receiving the second vaccination.) | 10 | 5
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.3) | 28.7 (6.2) | 34.7 (8.6) | 32.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 6 | 6 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 6 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 9 | 10 | 6 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of All Serious Adverse Events (SAEs) at Any Time During the Study
Time Frame: Day 1 post first vaccination to Day 180 post second vaccination
Population: One placebo subject was excluded from analysis (Did not receive vaccination).
Measure: Number; unit: Serious Adverse Event
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
Serious Adverse Event | 0 | 0 | 0

2. Primary Outcome: Occurrence of All Grade 3 Unsolicited Adverse Events (AEs) From First Vaccination Through Day 29 After the Second Vaccination
Time Frame: Through day 29 after the second vaccination
Population: One placebo subject was excluded from analysis (Did not receive vaccination).
Measure: Number; unit: Grade 3 Unsolicited Adverse Event
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
Grade 3 Unsolicited Adverse Event
  Related | 0 | 0 | 0
  Unrelated | 0 | 0 | 0

3. Primary Outcome: Occurrence of All Grade 3 Laboratory Toxicities From First Vaccination Through Day 15 After the Second Vaccination
Time Frame: Through day 15 after the second vaccination
Population: One placebo subject was excluded from analysis (Did not receive vaccination).
Measure: Number; unit: Grade 3 Laboratory Toxicities
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
Grade 3 Laboratory Toxicities
  Related | 0 | 0 | 0
  Unrelated | 0 | 0 | 1

4. Primary Outcome: Occurrence of Solicited Local AE and Reactogenicity Signs and Symptoms in the 7 Days After Each Vaccination
Time Frame: Through 7 days after each vaccination
Population: One subject in the low dose group withdrew prior to the second vaccination. One placebo subject was excluded from analysis (Did not receive vaccination).
Measure: Number; unit: Solicited Local Adverse Event
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
Solicited Local Adverse Event
  Any Local Symptom, Post-Dose 1, Day 0 | 0 | 1 | 0
  Any Local Symptom, Post-Dose 1, Day 1 | 1 | 4 | 0
  Any Local Symptom, Post-Dose 1, Day 2 | 0 | 3 | 0
  Any Local Symptom, Post-Dose 1, Day 3 | 0 | 0 | 0
  Any Local Symptom, Post-Dose 1, Day 4 | 0 | 0 | 0
  Any Local Symptom, Post-Dose 1, Day 5-7 | 0 | 0 | 0
  Any Local Symptom, Post-Dose 2, Day 0: number analyzed (Participants) | 9 | 10 | 5
  Any Local Symptom, Post-Dose 2, Day 0 | 0 | 0 | 0
  Any Local Symptom, Post-Dose 2, Day 1: number analyzed (Participants) | 9 | 10 | 5
  Any Local Symptom, Post-Dose 2, Day 1 | 3 | 3 | 0
  Any Local Symptom, Post-Dose 2, Day 2: number analyzed (Participants) | 9 | 10 | 5
  Any Local Symptom, Post-Dose 2, Day 2 | 1 | 1 | 1
  Any Local Symptom, Post-Dose 2, Day 3: number analyzed (Participants) | 9 | 10 | 5
  Any Local Symptom, Post-Dose 2, Day 3 | 1 | 0 | 0
  Any Local Symptom, Post-Dose 2, Day 4: number analyzed (Participants) | 9 | 10 | 5
  Any Local Symptom, Post-Dose 2, Day 4 | 1 | 0 | 0
  Any Local Symptom, Post-Dose 2, Day 5-7: number analyzed (Participants) | 9 | 10 | 5
  Any Local Symptom, Post-Dose 2, Day 5-7 | 0 | 0 | 0

5. Primary Outcome: Occurrence of Solicited Systemic AE and Reactogenicity Signs and Symptoms in the 7 Days After Each Vaccination
Time Frame: Through 7 days after each vaccination
Population: as for outcome 4
Measure: Number; unit: Solicited Systemic Adverse Event
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
Solicited Systemic Adverse Event
  Any Systemic Symptom, Post-Dose 1, Day 0 | 0 | 1 | 0
  Any Systemic Symptom, Post-Dose 1, Day 1 | 3 | 1 | 1
  Any Systemic Symptom, Post-Dose 1, Day 2 | 1 | 1 | 0
  Any Systemic Symptom, Post-Dose 1, Day 3 | 0 | 0 | 0
  Any Systemic Symptom, Post-Dose 1, Day 4 | 2 | 0 | 0
  Any Systemic Symptom, Post-Dose 1, Day 5-7 | 2 | 0 | 0
  Any Systemic Symptom, Post-Dose 2, Day 0: number analyzed (Participants) | 9 | 10 | 5
  Any Systemic Symptom, Post-Dose 2, Day 0 | 0 | 0 | 0
  Any Systemic Symptom, Post-Dose 2, Day 1: number analyzed (Participants) | 9 | 10 | 5
  Any Systemic Symptom, Post-Dose 2, Day 1 | 1 | 2 | 1
  Any Systemic Symptom, Post-Dose 2, Day 2: number analyzed (Participants) | 9 | 10 | 5
  Any Systemic Symptom, Post-Dose 2, Day 2 | 1 | 2 | 0
  Any Systemic Symptom, Post-Dose 2, Day 3: number analyzed (Participants) | 9 | 10 | 5
  Any Systemic Symptom, Post-Dose 2, Day 3 | 1 | 1 | 1
  Any Systemic Symptom, Post-Dose 2, Day 4: number analyzed (Participants) | 9 | 10 | 5
  Any Systemic Symptom, Post-Dose 2, Day 4 | 0 | 1 | 0
  Any Systemic Symptom, Post-Dose 2, Day 5-7: number analyzed (Participants) | 9 | 10 | 5
  Any Systemic Symptom, Post-Dose 2, Day 5-7 | 3 | 1 | 0

6. Primary Outcome: Occurrence of Any AE Through Day 29 After the Second Vaccination
Time Frame: Through day 29 after the second vaccination
Population: One placebo subject was excluded from analysis (Did not receive vaccination).
Measure: Number; unit: Adverse Event
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
Adverse Event
  At least one local solicited adverse event | 4 | 7 | 1
  At least one systemic solicited adverse event | 6 | 4 | 3
  At least one related unsolicited adverse event | 0 | 0 | 0
  At least one unrelated unsolicited adverse event | 6 | 7 | 5

7. Secondary Outcome: Percentage of Subjects Achieving Seroconversion (Greater Than or Equal to 1:10 in Plaque Reduction Neutralizing Titer [PRNT50] Titer) at Day 29 After First Vaccination and at Day 29 After Second Vaccination
Time Frame: At day 29 after first vaccination and at day 29 after second vaccination
Population: One low dose subject withdrew prior to the second vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
percentage of participants
  Day 29 Post Dose 1 | 10.0 [0.51 to 44.44] | 10.0 [0.51 to 44.44] | 0.0 [0.00 to 50.00]
  Day 29 Post Dose 2: number analyzed (Participants) | 9 | 10 | 5
  Day 29 Post Dose 2 | 22.2 [4.10 to 56.00] | 20.0 [3.68 to 55.56] | 0.0 [0.00 to 50.00]

8. Secondary Outcome: Geometric Mean Neutralizing Titers at Days 15 and 29 After First Vaccination and at Days 15, 29, 57, and 180 Following Second Vaccination
Time Frame: At days 15 and 29 after first vaccination and at days 15, 29, 57, and 180 following second vaccination
Population: One low dose subject withdrew prior to the second vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: PRNT50 GMT
Arm/Group | Low Dose | High Dose | Placebo
Number analyzed (Participants) | 10 | 10 | 5
PRNT50 GMT
  Day 15 Post Dose 1 | 5.00 [5 to 5] | 5.00 [5 to 5] | 5.00 [5 to 5]
  Day 29 Post Dose 1 | 5.74 [4.20 to 7.86] | 5.74 [4.20 to 7.86] | 5.00 [5 to 5]
  Day 15 Post Dose 2: number analyzed (Participants) | 9 | 10 | 5
  Day 15 Post Dose 2 | 7.35 [4.02 to 13.42] | 6.16 [4.40 to 8.60] | 5.00 [5 to 5]
  Day 29 Post Dose 2: number analyzed (Participants) | 9 | 10 | 5
  Day 29 Post Dose 2 | 7.35 [4.02 to 13.42] | 6.60 [4.09 to 10.65] | 5.00 [5 to 5]
  Day 57 Post Dose 2: number analyzed (Participants) | 9 | 10 | 5
  Day 57 Post Dose 2 | 6.80 [3.96 to 11.68] | 5.74 [4.20 to 7.86] | 5.00 [5 to 5]
  Day 180 Post Dose 2: number analyzed (Participants) | 9 | 10 | 5
  Day 180 Post Dose 2 | 5.83 [4.09 to 8.32] | 5.00 [5 to 5] | 5.00 [5 to 5]

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Low Dose | High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 6/10 | 7/10 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=10) | High Dose (N=10) | Placebo (N=5)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lipoedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Exposure to SARS- CoV-2 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT05172544/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT05172544/SAP_001.pdf
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT05172544/ICF_002.pdf